CLINICAL TRIAL: NCT04676958
Title: Effects of Vitamin K2 on Recovery From Muscle Damaging Exercise in Young and Older Adults
Brief Title: viTAmin K2 and rEcOVery From ExeRcise
Acronym: TAKEOVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: Kappa Bioscience (Unknown)
Responsible Party: Principal Investigator, Stuart Gray, Senior Lecturer, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 200190189
Record Dates: First submitted 2020-11-24; First posted 2020-12-21 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Inflammation; Oxidative Stress; Vitamin K; Exercise; Strength; Recovery
MeSH Terms: conditions — Inflammation; Motor Activity | interventions — Vitamin K 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 380 mg capsule/day micro-crystalline cellulose
  Interventions: Dietary Supplement: Micro-crystalline cellulose
- Vitamin K2 (Active Comparator): 380 mg capsule/day micro-crystalline cellulose including 240ug/day Vitamin K2
  Interventions: Dietary Supplement: Vitamin K2

INTERVENTIONS:
Dietary Supplement: Vitamin K2 — Vitamin K2
  Arms: Vitamin K2
Dietary Supplement: Micro-crystalline cellulose — Micro-crystalline cellulose
  Arms: Placebo

SUMMARY:
The aim of the current study, therefore, is to investigate the effects of vitamin K2 supplementation on the physiological responses to an acute bout of resistance exercise.

ELIGIBILITY:
Inclusion Criteria:

* Participant is able and willing to sign the Informed Consent From
* No plans to change lifestyle (activity and nutrition) during the study period
* Older group (n=40): 65 years of age or older.
* Younger group (n=40): Aged 18-40 years

Exclusion Criteria:

* Not currently, or in the last year, participating in more than 1h per week of vigorous aerobic physical activity or any resistance exercise
* BMI > 30 kg/m2
* diabetes
* severe cardiovascular disease
* seizure disorders
* liver disease
* uncontrolled hypertension (>150/90mmHg at baseline measurement)
* cancer or cancer that has been in remission <5 years
* ambulatory impairments which would limit ability to perform assessments of muscle function
* dementia
* currently taking Vitamin K2 supplements
* currently taking Vitamin K antagonists/anticoagulants (e.g. warfarin)
* current smoking
* history of drug abuse
* taking medication known to affect muscle (e.g. steroids).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Change in post exercise recovery of muscle strength | Change from baseline to 12 weeks
  Muscle strength (MVC) of the knee extensor muscles will be measured before and after (3h, 24h, 48h, 72h) an acute bout of resistance exercise

SECONDARY OUTCOMES:
Change in pain free range of motion during knee extension exercise | Change from baseline to 12 weeks
  The range of motion which is pain free will be measured during knee extension using a goniometer before and after (3h, 24h, 48h, 72h) an acute bout of resistance exercise
Change in post exercise recovery of functional abilities | Change from baseline to 12 weeks
  Time to complete 5 chair rises will be measured before and after (3h, 24h, 48h, 72h) an acute bout of resistance exercise
Change in post exercise recovery of sEMG activity | Change from baseline to 12 weeks
  Quadriceps muscle sEMG will be measured before and after (3h, 24h, 48h, 72h) an acute bout of resistance exercise
Change in post exercise interleukin-6 | Change from baseline to 12 weeks
  Circulating interleukin-6 will be measured before and after (3h, 24h, 48h, 72h) an acute bout of resistance exercise
Change in post exercise peroxiredoxin 3 redox state | Change from baseline to 12 weeks
  Circulating peroxiredoxin 3 redox state will be measured before and after (3h, 24h, 48h, 72h) an acute bout of resistance exercise
Change in vitamin K levels | Change from baseline to 12 weeks
  Vitamin K will be measured in baseline and 12 week samples
Change in Carboxylated Osteocalcin levels | Change from baseline to 12 weeks
  Carboxylated Osteocalcin will be measured in baseline and 12 week samples
Change in uncarboxylated Osteocalcin levels | Change from baseline to 12 weeks
  uncarboxylated Osteocalcin will be measured in baseline and 12 week samples
Change in carboxylated matrix gla-protein levels | Change from baseline to 12 weeks
  carboxylated matrix gla-protein will be measured in baseline and 12 week samples
Change in dephosphorylated-uncarboxylated matrix gla-protein levels | Change from baseline to 12 weeks
  dephosphorylated-uncarboxylated matrix gla-protein will be measured in baseline and 12 week samples
Change in post exercise F2 isoprostanes | Change from baseline to 12 weeks
  Circulating F2 isoprostanes will be measured before and after (3h, 24h, 48h, 72h) an acute bout of resistance exercise

OTHER OUTCOMES:
Change in lean mass | Change from baseline to 12 weeks
  Change in lean mass
Change in blood glucose | Change from baseline to 12 weeks
  Change in blood glucose
Change in blood lipids | Change from baseline to 12 weeks
  Change in blood lipids
Change in plasma insulin | Change from baseline to 12 weeks
  Change in plasma insulin
Change in fat mass | Change from baseline to 12 weeks
  Change in fat mass
Change in muscle thickness | Change from baseline to 12 weeks
  Change in muscle thickness
Change in exercise substrate utilisation | Change from baseline to 12 weeks
  Energy expenditure, carbodhydrate and fat oxidation during treadmill walking

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - University of Glasgow, Glasgow
  - Stuart Robert Gray, Glasgow

REFERENCES:
- [Derived] Lithgow H, Johnston L, Ho FK, Celis-Morales C, Cobley J, Raastad T, Hunter AM, Lees JS, Mark PB, Quinn TJ, Gray SR. Protocol for a randomised controlled trial to investigate the effects of vitamin K2 on recovery from muscle-damaging resistance exercise in young and older adults-the TAKEOVER study. Trials. 2022 Dec 20;23(1):1026. doi: 10.1186/s13063-022-06937-y. PMID 36539791